CLINICAL TRIAL: NCT06323096
Title: Разработка системы поддержки принятия клинических решений для тяжелых больных с политравмой
Brief Title: Development of Clinical Decision Support System for Severe Patients With Polytrauma
Status: Recruiting | Type: Observational
Sponsor: Semey State Medical University (Other)
Collaborators: Ministry of Science and Higher Education of the Republic of Kazakhstan (Other Government)
Responsible Party: Principal Investigator, Alexander Prokazyuk, MD, Anesthesiology and ICU specialist, Semey State Medical University
Other Study IDs: AR13067824
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Polytrauma
Keywords: severe polytrauma; clinical decision support system
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Polytrauma with SIRS: No intervention(s) to be administered.
- Polytrauma with Bloodloss: No intervention(s) to be administered.
- Polytrauma with ATC: No intervention(s) to be administered.
- Polytrauma with Pneumonia: No intervention(s) to be administered.

SUMMARY:
The goal of this observational study is to develop a Clinical Decision Support System for severe patients with polytrauma. The main questions it aims to answer are:

* Is it possible to predict the development of systemic inflammatory response syndrome for the next 24 h after admission?
* Is it possible to predict the development of blood loss >25% of blood volume for the next 24 h after admission?
* Is it possible to predict the development of acute traumatic coagulopathy for the next 24 h after admission?
* Is it possible to predict the development of pneumonia in polytrauma patients?
* Is it possible to predict the outcome in polytrauma patients?

No intervention is planned for this study.

DETAILED DESCRIPTION:
This study aimed to develop a Clinical Decision Support System for the management of severe polytrauma patients at the early inpatient care stage.

Scientific Hypothesis: It is assumed that the use of a clinical decision Support System at the stage of early inpatient care may reduce the mortality rate and adverse outcomes in severe patients with polytrauma.

Study setting The study is planned as a multicenter, non-interventional study, with participation from clinics providing inpatient trauma care for patients with polytrauma. The participating clinics will be selected based on their ability to provide access to a large and diverse population of patients with polytrauma. The research subgroup will be determined by clinics in compliance with the necessary ethical standards. The study will be conducted both retrospectively and prospectively, with data collection spanning a period of at least two years. Retrospective data will be collected from patients' medical records, including information on patient demographics, injury characteristics, diagnostic tests, and treatment modalities. Prospective data will be obtained through standardized patient interviews and clinical assessments, including patient-reported outcomes, clinical measures of physical and psychological functioning, and healthcare utilization. All participating clinics will be required to comply with the rules of medical ethics and deontology as well as local regulations governing access to personal data. In addition, researchers will be required to obtain informed consent from patients or their legal representatives before collecting any data for the study.

Obtained data:

Gender, Age, AIS code for every registered injury, NISS, Vitals on Admission (pulse rate, systolic and diastolic blood pressure, respiratory rate), Complete Blood Count on Admission (Red Blood Cells, Hematocrit, Hemoglobin, Platelets, White Blood Cells), biochemical analysis of blood on admission (total protein, total bilirubin, glucose, urea, creatinine), Blood Coagulation test (Activated Partial Thromboplastin Time, International Normalized Ratio, Fibrinogen), amount of total transfused blood and plasma packs, presence of complications (systemic inflammatory response syndrome, shock, severe hemorrhage [>25% of blood loss], acute traumatic coagulopathy, respiratory distress, pneumonia), length of stay in hospital, length of stay in the intensive care unit, and outcome at hospital discharge.

Additional Data Generation After the initial data were collected, additional fields will be created and calculated. These fields include the AIS field, which will be split into nine fields for each body region, with each field recording the square root of the sum of severity scores for that region; values for MCV, MCH, and MCHC, which will be calculated using the corresponding formulas; the "initial iron deficiency anemia" field, which will be calculated based on the initial MCV value; the "post-hemorrhagic anemia" field, which is calculated based on the initial hemoglobin level and relationship with initial iron deficiency anemia.

Informed Consent will be obtained by a research member who is an emergency/traumatology/ICU doctor, who was trained and explained to all the details of the current study. Consent will be obtained on patient admission to the hospital. Written Consent will be obtained from the patient or his/her legal representative if the patient is temporarily or completely disabled.

Recruitment will be started for every participating clinic separately during their recruitment periods, as defined by personal agreements. The main research clinic (Hospital of Emergency Aid, Semey, the Republic of Kazakhstan) has been participating in the recruitment process since December 1, 2020.

The reason for the recruitment end is the achievement of the minimum sample size by the research group or cancellation of participation in the trial.

The research group will collect a minimum sample size of data that will be used in the process of developing ML models. All the data were divided into training and test samples. Any record with less than 10% missing variables will have missing values imputed, whereas records with more than 10% missing variables will be excluded. Furthermore, additional data will be generated as outlined in the Eligibility Criteria section.

The selected features will be used to predict the following endpoints: the presence of complications (such as systemic inflammatory response syndrome, severe hemorrhage [>25% of blood loss], acute traumatic coagulopathy, respiratory distress, and pneumonia), and the outcome at hospital discharge.

All the developed models will be used for further CDSS development.

Confidentiality No identifiable patient information, such as names, IDs, phone numbers, emails, or addresses, will be collected. All information collected in accordance with the eligibility criteria will be transferred to trial participants via authorized access. After the study ends, any access not related to further work, such as statistical analysis or publications, will be blocked by the main researcher.

ELIGIBILITY:
Inclusion Criteria:

* Availability of informed consent, signed by the patient or his legal representative;
* Patients over 18 years of age;
* Expanded criteria of the new Berlin definition of polytrauma: patients who comply with three conditions:

  1. Presence of damage to one area of the body with an AIS score ≥3 points.
  2. Presence of damage to ≥2 areas of the body with an AIS score of ≥2.
  3. Presence of ≥1 physiological risk factors and/or primary hospitalization in the ICU.
* Completeness of the medical record in terms of laboratory and instrumental studies and protocol of therapeutic and surgical treatment.

Exclusion Criteria:

* Refusal to participate in the study at any stage.
* Death within one hour after hospitalization.
* Missing data.
* Patients who seek primary care 24 hours after injury.
* Patients requiring transfer between profiles and hospitals for implementation of rehabilitation or other stages of therapy.
* Patients with prematurely interrupted treatment.
* Trauma combined with suffocation, drowning, frostbite, electrical trauma, or chemical and/or thermal burns.
* Patients with pathological fractures.
* Pregnant women.
* Cases with predominantly severe craniocephalic (GCS <7 points) or spinal injury (deep paresis and plegias).

Min Age: 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: According to the World Health Organization (WHO forecast, by 2030 trauma is one of the five leading causes of death. In the Republic of Kazakhstan, road traffic injuries rank 7th among all causes of death (14.7 [the 10-year average is 16.9] per 100,000 population per year).
  Considering geographical and epidemiological factors, we chose two regional medical centers and the National Scientific Center of Traumatology and Orthopedics in the Republic of Kazakhstan, providing emergency medical care to patients with polytrauma (the serviced population is 610,000, 1,135,000, and 1,400,000 people, respectively).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Prediction of SIRS | By the end of January 2024
  Rate of SIRS prediction in the 24 h after admission using the developed CDSS.
Rate of ATC prediction in the 24 h after admission using the developed CDSS. | By the end of January 2024
  Rate of ATC prediction in the 24 h after admission using the developed CDSS.
Rate of hemorrage prediction in the 24 h after admission using the developed CDSS. | By the end of January 2024
  Rate of hemorrage prediction in the 24 h after admission using the developed CDSS.
Rate of pneumonia prediction using the developed CDSS. | By the end of January 2024
  Rate of pneumonia prediction within all period of admission using the developed CDSS.

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency Hospital, Semey, Abai, Kazakhstan

REFERENCES:
- [Derived] Prokazyuk A, Tlemissov A, Zhanaspayev M, Aubakirova S, Mussabekov A. Development and validation of a machine learning-based model to assess probability of systemic inflammatory response syndrome in patients with severe multiple traumas. BMC Med Inform Decis Mak. 2024 Aug 27;24(1):235. doi: 10.1186/s12911-024-02640-x. PMID 39192291